CLINICAL TRIAL: NCT04723225
Title: To Observe The Effectiveness Of Cat-Cow Yoga In The Pain Management Of Chronic Low Back Pain In Health Care Professionals
Brief Title: Effectiveness of Cat-Cow Yoga in Managing Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Responsible Party: Principal Investigator, Shamoon Noushad, Principal Investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PPL-CAT2020
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Chronic Low-back Pain
Keywords: Cat Cow Yoga; Yoga Therapy; Healthcare Providers; Substance P; Chronic low back pain; Cortisol; Beta Endorphins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Cat-Cow is one of the essential postures in yoga for its beneficial reasons. It is an alternate shift of posture from flexion of the back (rounded) to the extension of the back (arched). During each set of movement, inhalation and exhalation will be guided.
  Interventions: Other: Cat-Cow Yoga
- Control (No Intervention): In control intervention group usual care will be provided.

INTERVENTIONS:
Other: Cat-Cow Yoga — Cat-Cow is one of the essential postures in yoga for its beneficial reasons. It is an alternate shift of posture from flexion of the back (rounded) to the extension of the back (arched). During each set of movement, inhalation and exhalation will be guided
  Arms: Experimental

SUMMARY:
A randomized control trial is planned to investigate the effectiveness of Cat-Cow yoga as a treatment for chronic low back pain CLBP. An 12 weeks course of intervention will be provided to the candidates that will meet the eligibility criteria of the study. Substance P, beta endorphins and cortisol will be tested both the groups' pre and post treatment and then the difference from the baseline value will be determined.

DETAILED DESCRIPTION:
A randomized control trial will be conducted. Subjects who have passed the eligibility criteria will be asked for their consent to participate in the study. Then they will be chosen into their groups randomly. Every individual will have a fair chance to be selected in the test group in which they will receive the intervention, while the control group will receive 'usual care'. The outcomes of the study will be examined before the intervention and after the intervention with an interval of 12 weeks.

Subjects for this study will be enrolled from different Health care professionals of Karachi, Pakistan. Participants of the study will have diverse ethnicity, culture, socio-economic status etc. participants will be considered eligible for the study if the meet all the requirements of the inclusion criteria. Subjects will be invited and motivated for their participation in the study through advertisement on the notice board of their office. Those who have volunteered for the study will be provided with a consent form with detailed description of the study about its aims, duration and expected outcomes.

Interventions

The experimental intervention (Cat-Cow Yoga):

The cat-cow yoga therapy will be conducted in a conserved therapy center in Karachi. Session will start with a 10 minutes of warm-ups followed by 30 minutes of the therapy session in the afternoon three days a week (total 12 weeks).

The control intervention:

In control group, subjects will be given the usual care that if not vanishes the pain completely; will provide relief from the pain for the time being. Subjects in the control group will be asked to maintain a proper posture, take breaks during the work, remain active and to apply superficial heat if their pain exceeds their tolerance level.

ELIGIBILITY:
Inclusion Criteria:

Answer Yes to the following questions.

1. Have low back pain constantly or on most days for the last three months.
2. Have you seek care from health care provider due to back pain
3. Average pain intensity, assessed using the Numerical Pain Rating (NPR) scale over the past week ≥ 2 on a 0-10 numerical pain scale.
4. Roland Morris Disability Questionnaire score ≥ 4.
5. Fear Avoidance Beliefs Questionnaire (FABQ) work subscale score <19.

Exclusion Criteria:

* To be eligible for the study participants must not:

  * Have a personal history of the following neurological disorders: Alzheimer's, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Parkinson's, Stroke
  * Have a personal history of the following cardiorespiratory disorders: Congestive heart failure, Heart attack in past 24 months
  * Have a personal history of the following musculoskeletal disorders: Rheumatoid Arthritis, pathologic fractures of the spine, avascular necrosis or osteonecrosis, severe osteoarthritis. Including a history of spine surgery or a hip arthroplasty
  * Have active cancer
  * Be Blind
  * Report being pregnant, lactating, or that they anticipate becoming pregnant in the next 3-months
  * Have a body mass index greater than 35 kg/m2
  * Have clinical depression (i.e., subjects who score 24 or higher on the Center for Epidemiology Depression Scale).
  * Have used narcotics or muscle relaxants within 30 days prior to study enrollment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Pain Score | 3 Months
  It will assessed with the help of Numeric Pain Rating Scale. using a 0-10 scale, where 0 corresponds to "no pain" and 10 to "the greatest pain possible."
Extent of Disability | 3 Months
  It will be detected with the help of Oswestry Low Back Pain Disability Questionnaire. This index is considered a standard to assess low back functionality, it has a total of 10 sections, and for each section with a possible score 5. The percentage improvement is calculated through the total possible score x 100.

SECONDARY OUTCOMES:
Substance P | 3 Months
  Changes in the levels of Substance P will be observed during the span of the study in test and control groups.
Beta Endorphins | 3 Months
  Changes in the levels of beta endorphins will be observed during the span of the study in test and control groups.
Stress Score | 3 Months
  Physical stress of the participants will be evaluated with Sadaf Stress Scale (SSS) before and after the therapy in both the groups.
Cortisol | 3 Months
  Changes in the levels of Cortisol will be observed during the span of the study in test and control groups.
Quality of Life Score | 3 Months
  This measure will be evaluated from baseline to post intervention with the help of World Health organization Quality of Life (WHOQOL) Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Koohi Goth Women Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noushad S, Ansari B, Ahmed S. Effect of nature-based physical activity on post-traumatic growth among healthcare providers with post-traumatic stress. Stress Health. 2022 Oct;38(4):813-826. doi: 10.1002/smi.3135. Epub 2022 Feb 26. PMID 35191173
- [Background] Noushad S, Ahmed S, Ansari B, Mustafa UH, Saleem Y, Hazrat H. Physiological biomarkers of chronic stress: A systematic review. Int J Health Sci (Qassim). 2021 Sep-Oct;15(5):46-59. PMID 34548863
- [Result] Holtzman S, Beggs RT. Yoga for chronic low back pain: a meta-analysis of randomized controlled trials. Pain Res Manag. 2013 Sep-Oct;18(5):267-72. doi: 10.1155/2013/105919. Epub 2013 Jul 26. PMID 23894731
- [Result] Cramer H, Lauche R, Haller H, Dobos G. A systematic review and meta-analysis of yoga for low back pain. Clin J Pain. 2013 May;29(5):450-60. doi: 10.1097/AJP.0b013e31825e1492. PMID 23246998
- [Result] Goode AP, Coeytaux RR, McDuffie J, Duan-Porter W, Sharma P, Mennella H, Nagi A, Williams JW Jr. An evidence map of yoga for low back pain. Complement Ther Med. 2016 Apr;25:170-7. doi: 10.1016/j.ctim.2016.02.016. Epub 2016 Mar 3. PMID 27062965
- [Result] Zhu F, Zhang M, Wang D, Hong Q, Zeng C, Chen W. Yoga compared to non-exercise or physical therapy exercise on pain, disability, and quality of life for patients with chronic low back pain: A systematic review and meta-analysis of randomized controlled trials. PLoS One. 2020 Sep 1;15(9):e0238544. doi: 10.1371/journal.pone.0238544. eCollection 2020. PMID 32870936
- [Result] Alleva J, Hudgins T, Belous J, Kristin Origenes A. Chronic low back pain. Dis Mon. 2016 Sep;62(9):330-3. doi: 10.1016/j.disamonth.2016.05.012. Epub 2016 Jun 22. No abstract available. PMID 27344193
- [Result] Sanzarello I, Merlini L, Rosa MA, Perrone M, Frugiuele J, Borghi R, Faldini C. Central sensitization in chronic low back pain: A narrative review. J Back Musculoskelet Rehabil. 2016 Nov 21;29(4):625-633. doi: 10.3233/BMR-160685. PMID 27062464
- [Result] Patrick N, Emanski E, Knaub MA. Acute and chronic low back pain. Med Clin North Am. 2014 Jul;98(4):777-89, xii. doi: 10.1016/j.mcna.2014.03.005. PMID 24994051
- [Result] Zieglgansberger W. Substance P and pain chronicity. Cell Tissue Res. 2019 Jan;375(1):227-241. doi: 10.1007/s00441-018-2922-y. Epub 2018 Oct 3. PMID 30284083
- [Result] Kallman TF, Ghafouri B, Backryd E. Salivary beta-endorphin and substance P are not biomarkers of neuropathic chronic pain propensity. Heliyon. 2018 Aug 3;4(8):e00718. doi: 10.1016/j.heliyon.2018.e00718. eCollection 2018 Aug. PMID 30116793
- [Result] Lisowska B, Lisowski A, Siewruk K. Substance P and Chronic Pain in Patients with Chronic Inflammation of Connective Tissue. PLoS One. 2015 Oct 7;10(10):e0139206. doi: 10.1371/journal.pone.0139206. eCollection 2015. PMID 26444559
- [Result] Veening JG, Barendregt HP. The effects of beta-endorphin: state change modification. Fluids Barriers CNS. 2015 Jan 29;12:3. doi: 10.1186/2045-8118-12-3. PMID 25879522